CLINICAL TRIAL: NCT02890628
Title: Perceptions and Experiences of Teenage Pregnancies in Refugee and Migrant Adolescents on the Thai-Myanmar Border
Brief Title: Teenage Pregnancies in Refugee and Migrant Adolescents on the Thai-Myanmar Border
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: SMRU 1602
Record Dates: First submitted 2016-07-13; First posted 2016-09-07 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Teenage Pregnancy
Keywords: Thai-Myanmar border

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- pregnant/post-natal adolescents (<20 years): 12-24 individual with pregnant or postnatal adolescent girls (<20 years) will be interviewed.
- non-pregnant female adolescents (<20 years): 1 Focus group discussion of 6-10 non-pregnant female adolescents (<20 years)
- male adolescents (<20 year): 1 Focus group discussion of 6-10 adolescent men (<20 years)
- SMRU health staff of antenatal clinics (ANC): 1 Focus group discussion of 6-10 Shoklo Malaria Research Unit antenatal clinic staff

SUMMARY:
This study is to explore perceptions, experiences, beliefs and knowledge around teenage pregnancy, motherhood, sexual and reproductive health, family planning and support structures adolescent refugees and migrants and to identify demographic, social and medical characteristics of study participants.

DETAILED DESCRIPTION:
The study will be conducted as follows:

* 12-24 individual interviews with pregnant or postnatal adolescent girls (<20 years);
* 1 Focus group discussion of 6-10 non-pregnant female adolescents (<20 years);
* 1 Focus group discussion of 6-10 adolescent men (<20 years);
* 1 Focus group discussion of 6-10 Shoklo malaria research unit antenatal care staff;

Interviews and focus group discussion will be conducted with study participants who agree to participate in discussions about teenage pregnancy and motherhood, sexual and reproductive health. In-depth interviews and focus group discussion will be conducted in private meeting rooms in proximity to the antenatal clinic waiting areas. In-depth interviews and Focus group discussion will be co-facilitated by the principal investigator and a trained counsellor/midwife fluent in Karen, Burmese and English. Focus group discussion will be run separately for Burmese- and Karen-speaking participants and participants will be separated by subgroup. Focus group discussion will include 6-10 participants per group and for each focus group discussion to last between 45-60 minutes. Individual in-depth interviews will last approximately 60 minutes each.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for adolescent mothers (subgroup 1) are:

* Aged 12 - <20 years
* Females
* Migrant or refugee status
* Myanmar nationality
* Any trimester of pregnancy or up to 12 month post partum
* Able and willing to participate and give informed consent

Inclusion criteria for non-pregnant female adolescents (subgroup 2) are:

* Aged <20 years
* Females
* Migrant or refugee status
* Myanmar nationality
* No past or current pregnancy
* Able and willing to participate and give informed consent

Inclusion criteria for adolescent men (subgroup 3) are:

* Aged <20 years
* Males
* Migrant or refugee status
* Myanmar nationality
* Able and willing to participate and give informed consent

Inclusion criteria for health staff (subgroup 4) are:

* No age restrictions
* Females or males
* Migrant, refugee or non-migrant status
* Any nationality
* Able and willing to participate and give informed consent

Exclusion Criteria:

* Any participant who is deemed by the researchers or health staff to be acutely physically or mentally unwell will be excluded.
* Participants who do not meet the age requirements, migration status or nationality requirements

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The participant will be adolescent mothers and non-pregnant adolescent aged 12 - <20 years, adolescent men aged < 20 years and ANC staff.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2016-09; Primary Completion 2016-09-21 (Actual); Study Completion 2016-09-21 (Actual)

PRIMARY OUTCOMES:
Thematic summary of adolescents' perceptions, experiences and beliefs in teenage pregnancy, motherhood, sexual and reproductive health, family planning and support structures adolescent refugees and migrants | up to 1 year
Descriptive summary of demographic, social and medical characteristics of study participants | up to 1 year

SECONDARY OUTCOMES:
Summary of antenatal clinic staff perceptions | up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Shoklo Malaria Research Unit, Mae Sot, Changwat Tak, Thailand

IPD SHARING:
Plan to Share IPD: Yes